CLINICAL TRIAL: NCT05690750
Title: Gastric Antral Vascular Ectasia in Patients With Cirrhosis: Risk-factors and Associations.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-54
Record Dates: First submitted 2023-01-02; First posted 2023-01-19 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Gastric Antral Vascular Ectasia; Liver Cirrhosis
MeSH Terms: conditions — Gastric Antral Vascular Ectasia; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Cirrhosis with GAVE
  Interventions: Other: No intervention
- Control: Cirrhosis without GAVE
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention as this is an observational study.

SUMMARY:
We will evaluate all out-patients and in-patients with cirrhosis, who undergo upper gastrointestinal endoscopy (EGD) in the Department of Hepatology, Institute of Liver and Biliary Sciences (ILBS), for inclusion. Patients with cirrhosis, with age >18-years, who have characteristic findings of GAVE on endoscopy will be included in this study. Their clinical and biochemical features, and endoscopy findings will be compared with a gender and age-matched control group of cirrhosis without GAVE. This observational, case-control study will aim to define the predictors of GAVE in patients with cirrhosis.

DETAILED DESCRIPTION:
Primary Objective: To study whether GAVE is more prevalent among patients with cirrhosis who have diabetes mellitus, compared to cirrhotic patients without diabetes.

- Secondary objectives:

1. Relationship of etiology of cirrhosis with occurrence of GAVE.
2. Relationship of severity of cirrhosis (CTP score and MELD score), with GAVE.
3. Features of metabolic syndrome among cirrhotic patients with GAVE.
4. Variceal grade and previous endotherapy with occurrence of GAVE among patients with cirrhosis.
5. Prevalence of proximal gastric vascular ectasias among cirrhotic patients with GAVE.

   (b) Methodology:
   * Study population:

   All out-patients and in-patients who undergo upper gastrointestinal endoscopy (EGD) in the Department of Hepatology, Institute of Liver and Biliary Sciences (ILBS), will be evaluated for inclusion. Diagnosis of cirrhosis will be based on a combination of imaging features, liver biopsy, elastography measurements, and signs of portal hypertension.

   We will include patients with cirrhosis with age >18-years, who have characteristic findings of GAVE on endoscopy in this study.

   - Study design:

   Case-control, observational study.
   * Study period:

     3-months.
   * Sample size with justification:

   There are three existing studies which have shown an association of diabetes mellitus (DM) with occurrence of GAVE [Fouad M. JGH Open 2021; Smith E. Am J Med 2016; Cleach AL. Canadian Liver Journal 2019]. The prevalence of DM among patients with and without GAVE ranged from 50%-64%, and 24.2% to 29.3%, respectively, in these three studies.

   Assuming a prevalence of DM of 50% among cirrhosis patients with GAVE, and 25% prevalence of DM among cirrhotic patients without GAVE, we will need 44 cases (and 88 controls) to detect a difference with power of 80% and significance level of 0.05, using the test of independent proportions. We plan to include 50 cases and 100 controls in this study.

   - Intervention: None.

   - Monitoring and assessment: Not applicable.
   * Statistical Analysis:

   Patients with GAVE will be matched in a 1:2 ratio to controls without GAVE, based on age (±5 years), gender, and timing of diagnostic EGD (±1 year). Comparisons will be performed using Chi-square tests or Fisher exact tests for categorical variables, and t tests, Wilcoxon rank-sum tests or signed rank tests for continuous variables as appropriate.

   Univariate and multivariate, case and control matched conditional logistic regression models will be utilized to evaluate potential associations between specific risk factors and the diagnosis of GAVE. A p≤0.05 decision rule is established a priori as the null hypothesis rejection rule for all comparisons.

   - Adverse effects:

   No intervention planned, hence no adverse effects anticipated.

   - Stopping rule of study:

   Not applicable.

   (c) Expected outcome of the project:

   Elucidation of the predictors of GAVE in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

- All patients with cirrhosis, with age >18-years, who have characteristic findings of GAVE on endoscopy.

Exclusion Criteria:

1. Active upper GI bleeding preventing adequate mucosal evaluation.
2. Patients unable or unwilling to give informed consent.
3. Endoscopic treatment of GAVE in past one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All out-patients and in-patients who undergo upper gastrointestinal endoscopy (EGD) in the Department of Hepatology, Institute of Liver and Biliary Sciences (ILBS), will be evaluated for inclusion. Diagnosis of cirrhosis will be based on a combination of imaging features, liver biopsy, elastography measurements, and signs of portal hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gastric antral vascular ectasia (GAVE) among cirrhotic patients with diabetes mellitus (fasting blood sugar>126mg/dL, and/or HbA1c >6.5%), compared to cirrhotic patients without diabetes. | 3 months

SECONDARY OUTCOMES:
Comparison of Model for End-Stage Liver Disease (MELD) scores (on a scale of 6-40) of cirrhotic patients with GAVE and cirrhotic patients without GAVE. | 3 months
Comparison of Child Turcotte Pugh (CTP) scores (on a scale of 5-15) of cirrhotic patients with GAVE and cirrhotic patients without GAVE. | 3 months
Grade of esophageal varices among cirrhotic patients with GAVE, compared to cirrhotic patients without GAVE. | 3 months
Prevalence of proximal gastric vascular ectasias among cirrhotic patients with GAVE. | 3 months
Comparison of the number of features of metabolic syndrome among cirrhotic patients with GAVE and cirrhotic patients without GAVE. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided